CLINICAL TRIAL: NCT00598390
Title: PET Test/Retest Brain Imaging of Cannabinoid CB1 Receptors Using [11C]MePPEP
Brief Title: PET Imaging of Cannabinoid CB1 Receptors Using [11C]MePPEP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 080048; 08-M-0048
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2013-01-22

CONDITIONS: Healthy
Keywords: Cannabinoid; CB1 Receptor; Brain Imaging; PET Imaging; [11C]MePPEP; Healthy Volunteer; HV
MeSH Terms: interventions — 5-(3-methoxyphenyl)-3-(1-phenylethylamino)-1-(4-trifluoromethylphenyl)pyrrolidin-2-one

INTERVENTIONS:
Drug: [11C]MePPEP

SUMMARY:
The purpose of this protocol is to measure brain CB1 receptors in the hope to better understand how they work, so that one day we can understand how the CB1 receptors are involved in psychiatric, neurological, and behavioral disorders.

DETAILED DESCRIPTION:
MePPEP is a ligand that is highly selective for the cannabinoid type 1 (CB1) receptor. This receptor is considered the most common G-coupled protein receptor in the brain (Pacher et al., 2006). The CB1 receptor is the site of action of Delta-9-tetrahydrocannbinol (THC), the active compound in marijuana, and is found primarily on the presynaptic terminals of dopaminergic, glutamatergic, GABAergic neurons (Howlett et al., 2002). The function of the CB1 receptor is not entirely clear; however, it has been implicated in several neurological and psychiatric disorders, and a selective inverse agonist, rimonabant, is currently in use in Europe for the treatment of obesity (Van Gaal et al., 2005). [11C]MePPEP was developed to enhance our understanding of the in vivo characteristics of the CB1 receptor (e.g., receptor density and receptor occupancy with pharmaceuticals).

The purpose of this protocol is to establish an accurate method to measure CB1 receptor levels in brain by performing test/retest brain imaging studies. The results of this overall study are required to apply this PET ligand in various neurological and psychiatric disorders in the future.

ELIGIBILITY:
* INCLUSION CRITERIA:

<TAB>

All subjects must be healthy and aged 18 65 years, with history/physical exam, ECG, and laboratory tests within one year of the PET scan. The volunteer must sign an informed consent form.

EXCLUSION CRITERIA:

* Current psychiatric illness, substance abuse including marijuana use, or severe systemic disease based on history and physical exam.
* Laboratory tests with clinically significant abnormalities or positive urine toxicology screen.
* Prior participation in other research protocols in the last year such that radiation exposure would exceed the annual limits.
* Pregnancy and breast feeding.
* Claustrophobia.
* Presence of ferromagnetic metal in the body or heart pacemaker.
* Positive HIV test.
* Employee of the investigative site or an immediate family member of an employee of the investigative site. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Employee of Eli Lilly and Company.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-01-08; Primary Completion 2013-01-22 (Actual); Study Completion 2013-01-22 (Actual)

PRIMARY OUTCOMES:
Reproducibility of novel PET tracer for CB1 in brain imaging.

SECONDARY OUTCOMES:
Distribution and variance of CB1 receptors in the brain of healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abi-Dargham A, Gandelman M, Zoghbi SS, Laruelle M, Baldwin RM, Randall P, Zea-Ponce Y, Charney DS, Hoffer PB, Innis RB. Reproducibility of SPECT measurement of benzodiazepine receptors in human brain with iodine-123-iomazenil. J Nucl Med. 1995 Feb;36(2):167-75. PMID 7830108
- [Background] Burger C, Buck A. Requirements and implementation of a flexible kinetic modeling tool. J Nucl Med. 1997 Nov;38(11):1818-23. PMID 9374364
- [Background] Carson RE, Huang SC, Green MV. Weighted integration method for local cerebral blood flow measurements with positron emission tomography. J Cereb Blood Flow Metab. 1986 Apr;6(2):245-58. doi: 10.1038/jcbfm.1986.38. PMID 3485644